CLINICAL TRIAL: NCT02712476
Title: Comparison of Mannitol Alone Versus Different Doses of Mannitol in Combination With Furosemide on Brain Relaxation in Supratentorial Mass Resection Surgery
Brief Title: Brain Relaxation With Mannitol and Furosemide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Eren Fatma Akcil, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cerrahpasa Neuroanesthesia
Record Dates: First submitted 2016-03-01; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Brain Tumors
Keywords: Mannitol; Furosemid; Brain Relaxation
MeSH Terms: conditions — Brain Neoplasms | interventions — Mannitol; Furosemide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol,furosemide (Active Comparator): Mannitol 0.5mg/kg and furosemide 0.5mg/kg IV is compared with mannitol 1mg/kg and furosemide 0.5mg/kg
  Interventions: Drug: mannitol; Drug: Furosemide
- Mannitol, placebo (Placebo Comparator): Mannitol 0.5mg/kg and placebo is compared with mannitol+forosemide
  Interventions: Drug: mannitol; Drug: placebo

INTERVENTIONS:
Drug: mannitol — This drug is in our routine use of neuroanesthesia, are given in peroperatifyl brain relaxation
Drug: Furosemide — This drug is can be used alone or with mannitol for brain relaxation
  Other Names: Lasix
  Arms: Mannitol,furosemide
Drug: placebo — mannitol alone is compared with placebo
  Arms: Mannitol, placebo

SUMMARY:
Although mannitol is used for brain relaxation during neurosurgery and in the treatment of raised intracranial pressure; there is not a consensus on its safe and effective dose, the duration of its administration and its use in combination with loop diuretics. This study aimed to compare the effects of the mannitol alone and in combination with furosemide in different doses, on the brain relaxation, electrolyte, lactate levels of the blood, peroperative fluid balance and the volume of the urine in supratentorial mass resection surgeries.

This prospective, randomized, double blind, placebo controlled study included fifty one patients (ASA I-III) scheduled for elective supratentorial mass resection surgery. The patients were randomized into three groups for investigation of the effects of mannitol alone and in combination with furosemide in different doses. Blood sodium, potassium, chlorine, lactate, urine and osmolarity levels were recorded. The brain relaxation score (BRS) was evaluated twice by the surgeon using a 4 point scale (1=very good, 2=good, 3=bad, 4=very bad); at dura opening, and 30 minutes after the administration of the study drug.

DETAILED DESCRIPTION:
After obtaining approval from the ethics committee and informed consent, a total of 51 patients aged 20-70 years, conscious and American Society of Anesthesiologists (ASA) class I-III, who had intracranial shift and who were scheduled for supratentorial mass resection under elective conditions, were included in the present prospective, randomized, double-blind and placebo-controlled study. Patients with decompensated heart failure, kidney insufficiency, diabetes insipidus, electrolyte imbalance and who are unconscious were excluded from the study.

Drug doses were determined based on the ideal body weight (IBW) or adjusted body weight (ABW) if the real body weight was 30 percent higher than the calculated ideal weight.

After premedication with midazolam (0.03 mg.kg-1) (Dormicum®, Roche, Basel, Switzerland), the patients were moved to the operating room and placed under continuous monitoring with electrocardiography (ECG), non-invasive blood pressure measurement and peripheral oxygen saturation. Intravenous (IV) bolus doses of propofol (2 mg.kg-1) (Propofol®, Fresenius Kabi, Homburg, Germany) rocuronium (0.6 mg.kg-1) (Curon®, Mustafa Nevzat, Istanbul, Turkey), remifentanil infusion (0.15 µg.kg-1) (Ultiva®, Glaxo Smith Kline, London, UK) and 0.7 FiO2 oxygen-air were used in the induction of anesthesia, while remifentanil (0.15 µg.kg-1) (Ultiva®, Glaxo Smith Kline, London, UK), rocuronium (0.03 mg.kg-1) (Curon®, Mustafa Nevzat, Istanbul, Turkey) infusions, and 0.5-1 MAC sevoflurane (Sevorane®, Abbvie, North Chicago, USA) in a mixture of 0.4 FiO2 oxygen-air were used in the maintenance. A nasogastric tube was inserted into each patient after intubation, and invasive blood pressure monitoring was continued with arterial cannulation, while urine output was monitored by inserting a foley urinary catheter. The body temperature was measured by urinary catheter. In the IV fluid management; balanced fluids were administered (Isolayte-S® , Eczacıbaşı Baxter, Istanbul, Turkey) for maintenance and replacement, colloids and blood products were also administered in the case of bleeding. At the time of wound closure tramadol 100 mg (Contramal®, Abdi İbrahim, Istanbul, Turkey) and ondansetron 8 mg IV (Zofer®, Glaxo Smith Kline, London, UK) were administered. At the end of the operation, decurarization was carried out through the administration of atropine (0.01 mg.kg-1) (Atropine sülfat®, Galen, Istanbul, Turkey) and neostigmine (0.02 mg.kg-1) (Neostigmine®, Adeka, Samsun, Turkey).

The patients were randomized into 3 groups using a closed envelope method, group 1; mannitol 0.5 g.kg-1 and furosemide 0.5 mg.kg-1 (G1), group 2; mannitol 1 g.kg-1 and furosemide 0.5 mg.kg-1 (G2) and group 3; mannitol 0.5 g.kg-1 and placebo (G3). All medications were prepared by a single nurse in 100 mL of a 0.9 percent isotonic saline solution. After head fixation, all patients were administered with mannitol (over 20 minutes) and the study drug. Arterial blood gas (ABG) analysis (Cobas b 221 blood gas analyzer, Roche®, Basel, Switzerland) was made at 30 minute intervals in the first 2 hour and then again in the 6th, 12th and 24th hours after study drug administration. Blood sodium, potassium, chlorine, lactate levels and urine output were recorded in each intervals. Blood osmolarity measured levels were recorded before the study drug administration and 2nd hours. The brain relaxation score (BRS) was evaluated twice by the surgical team using a 4 point scale (1= very good, 2= good, 3= bad, 4= very bad); first, at the time of dura opening, and second, 30 minutes after the administration of the study drug.

All patients were extubated at the end of the surgery and followed in the neurosurgical-intensive care unit (NICU) for 24 hours postoperatively.

The surgery type was recorded. The volume of peroperative blood loss, transfused blood products, the volume of the given peroperative IV fluids and fluid balance were also recorded.

Statistical analysis:

On the basis of previous study (10) and the assumption that a difference of 1 unit on BRS from 1 to 4 in brain relaxation is clinically relevant, setting α equal to 0.05 and β equal to 0.9, we calculated a sample size of 15 patients per group. To compensate for dropouts, the study included 51 patients.

Statistical analysis was performed using SPSS (Statistical Package for Social Sciences) for Windows 21.0. Differences between the groups were analysed by using one-way analysis of variance (ANOVA) with the post-hoc Tukey analysis. The differences in ASA, gender and BRS between groups were analyzed by using Pearson chi-square test. Differences within groups in electrolyte and lactate levels, osmolarity and BRS were analyzed by repeated measures of ANOVA with the post-hoc Bonferroni correction test. Values of p ≤ 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial shift
* Scheduled for supratentorial mass resection under elective conditions

Exclusion Criteria:

* Decompensated heart failure
* kidney insufficiency
* Diabetes insipidus,
* Electrolyte imbalance and
* Who are unconscious

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
brain relaxation score | Change in brain relaxation in 30 minutes after drug administration
  evaluated by surgical team using 4 point scale (1= very good, 2= good, 3= bad, 4= very bad)

SECONDARY OUTCOMES:
Blood sodium levels (mEq/L) | change in 30 minute intervals in the first 2 hour and then again in the 6th, 12th and 24th hours after study drug administration
Blood potassium levels (mEq/L) | change in 30 minute intervals in the first 2 hour and then again in the 6th, 12th and 24th hours after study drug administration
Blood chlorine levels (mEq/L) | change in 30 minute intervals in the first 2 hour and then again in the 6th, 12th and 24th hours after study drug administration
Blood lactate levels (mmol/L) | change in 30 minute intervals in the first 2 hour and then again in the 6th, 12th and 24th hours after study drug administration
24 hours diuresis (mL) | change in 24th hours after study drug administration
Fluid balance during operation (mL) | Change in balance during operation time

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vialet R, Leone M, Albanese J, Martin C. Calculated serum osmolality can lead to a systematic bias compared to direct measurement. J Neurosurg Anesthesiol. 2005 Apr;17(2):106-9. doi: 10.1097/01.ana.0000163200.48483.56. PMID 15840998
- [Result] Bebawy JF, Ramaiah VK, Zeeni C, Hemmer LB, Koht A, Gupta DK. The effect of furosemide on intravascular volume status and electrolytes in patients receiving mannitol: an intraoperative safety analysis. J Neurosurg Anesthesiol. 2013 Jan;25(1):51-4. doi: 10.1097/ANA.0b013e318269c335. PMID 23237936
- [Result] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. XV. Steroids. J Neurotrauma. 2007;24 Suppl 1:S91-5. doi: 10.1089/neu.2007.9981. No abstract available. PMID 17511554
- [Result] Li Q, Chen H, Hao JJ, Yin NN, Xu M, Zhou JX. Agreement of measured and calculated serum osmolality during the infusion of mannitol or hypertonic saline in patients after craniotomy: a prospective, double-blinded, randomised controlled trial. BMC Anesthesiol. 2015 Oct 7;15:138. doi: 10.1186/s12871-015-0119-4. PMID 26445777
- [Result] Manninen PH, Lam AM, Gelb AW, Brown SC. The effect of high-dose mannitol on serum and urine electrolytes and osmolality in neurosurgical patients. Can J Anaesth. 1987 Sep;34(5):442-6. doi: 10.1007/BF03014345. PMID 3117392
- [Result] Pollay M, Fullenwider C, Roberts PA, Stevens FA. Effect of mannitol and furosemide on blood-brain osmotic gradient and intracranial pressure. J Neurosurg. 1983 Dec;59(6):945-50. doi: 10.3171/jns.1983.59.6.0945. PMID 6415245
- [Result] Procaccio F, Stocchetti N, Citerio G, Berardino M, Beretta L, Della Corte F, D'Avella D, Brambilla GL, Delfini R, Servadei F, Tomei G. Guidelines for the treatment of adults with severe head trauma (part II). Criteria for medical treatment. J Neurosurg Sci. 2000 Mar;44(1):11-8. PMID 10961491
- [Result] Procaccio F, Stocchetti N, Citerio G, Berardino M, Beretta L, Della Corte F, D'Avella D, Brambilla GL, Delfini R, Servadei F, Tomei G. Guidelines for the treatment of adults with severe head trauma (part I). Initial assessment; evaluation and pre-hospital treatment; current criteria for hospital admission; systemic and cerebral monitoring. J Neurosurg Sci. 2000 Mar;44(1):1-10. PMID 10961490
- [Result] Quentin C, Charbonneau S, Moumdjian R, Lallo A, Bouthilier A, Fournier-Gosselin MP, Bojanowski M, Ruel M, Sylvestre MP, Girard F. A comparison of two doses of mannitol on brain relaxation during supratentorial brain tumor craniotomy: a randomized trial. Anesth Analg. 2013 Apr;116(4):862-8. doi: 10.1213/ANE.0b013e318282dc70. Epub 2013 Jan 25. PMID 23354336
- [Result] Rozet I, Tontisirin N, Muangman S, Vavilala MS, Souter MJ, Lee LA, Kincaid MS, Britz GW, Lam AM. Effect of equiosmolar solutions of mannitol versus hypertonic saline on intraoperative brain relaxation and electrolyte balance. Anesthesiology. 2007 Nov;107(5):697-704. doi: 10.1097/01.anes.0000286980.92759.94. PMID 18073543
- [Result] Schettini A, Stahurski B, Young HF. Osmotic and osmotic-loop diuresis in brain surgery. Effects on plasma and CSF electrolytes and ion excretion. J Neurosurg. 1982 May;56(5):679-84. doi: 10.3171/jns.1982.56.5.0679. PMID 6802937
- [Result] Thenuwara K, Todd MM, Brian JE Jr. Effect of mannitol and furosemide on plasma osmolality and brain water. Anesthesiology. 2002 Feb;96(2):416-21. doi: 10.1097/00000542-200202000-00029. PMID 11818776
- [Result] Todd MM, Cutkomp J, Brian JE. Influence of mannitol and furosemide, alone and in combination, on brain water content after fluid percussion injury. Anesthesiology. 2006 Dec;105(6):1176-81. doi: 10.1097/00000542-200612000-00017. PMID 17122580
- [Derived] Akcil EF, Dilmen OK, Karabulut ES, Koksal SS, Altindas F, Tunali Y. Effective and safe mannitol administration in patients undergoing supratentorial tumor surgery: A prospective, randomized and double blind study. Clin Neurol Neurosurg. 2017 Aug;159:55-61. doi: 10.1016/j.clineuro.2017.05.018. Epub 2017 May 15. PMID 28544917
- See also: test link — http://www.ncbi.nlm.nih.gov/pubmed